CLINICAL TRIAL: NCT00772447
Title: A Phase 3, Multicentre, Randomised, Investigator-blinded, Parallel-groupStudy of the Safety and Efficacy of Intravenous Daptomycin (Cubicin®)Compared With That of Comparator (Vancomycin or Vancomycin Followed by Semi-synthetic Penicillin-cloxacillin) in the Treatment of Chinese Subjects With cSSSI
Brief Title: China Registration Study in Patients With Skin Infections
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D1790C00003
Record Dates: First submitted 2008-10-09; First posted 2008-10-15 (Estimated); Results first posted 2015-03-09 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-02

CONDITIONS: Skin Diseases; Infectious
Keywords: Skin Infections; Complicated Bacterial Skin and Skin Structure Infection due to Gram-positive Pathogens
MeSH Terms: conditions — Skin Diseases; Communicable Diseases; Cellulitis | interventions — Daptomycin; Vancomycin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AZ drug (Experimental): Daptomycin
  Interventions: Drug: Daptomycin
- Comparator (Active Comparator): Vancomycin or Vancomycin Followed by Semi-synthetic Penicillin-Cloxacillin
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Daptomycin — 4mg/kg IV ; Q 24 hr (once every 24 hours)
  Other Names: Cubicin®
  Arms: AZ drug
Drug: Vancomycin — Vancomycin - 1g per 12 hrs, for 7-14 days
  Or switch to
  Vancomycin Followed by Semi-synthetic Penicillin-Cloxacillin:
  - 1 g every 6 hours or 2 g every 8 hours
  Arms: Comparator

SUMMARY:
The objectives of this study is to evaluate the Safety and Efficacy of Intravenous Daptomycin (Cubicin®)Compared with that of Comparator (Vancomycin or Vancomycin Followed by Semi-synthetic Penicillin-cloxacillin) in the Treatment of Chinese Subjects with Complicated Bacterial Skin and Skin Structure Infection due to Gram-Positive Pathogens.

ELIGIBILITY:
Inclusion Criteria:

* Provision of inform consent
* A diagnosis of of complicated skin and skin structure infection known or suspected to be due to Gram-positive bacteria
* Diagnosis of bacterial skin and skin structure infection in the presence of some complicating factor, including infections involving deeper soft tissue or requiring surgical intervention, a pre-existing lesion or underlying condition affect healing

Exclusion Criteria:

* Subjects known to have any bloodstream infection (including bloodstream infection caused by S. aureus). Subjects whose baseline blood cultures are positive for any clinically pathogenic organism ( including S. aureus ) should be discontinued from study
* Minor or superficial skin infections, Infected "decubitus"ulcer, Perirectal abscess, Hidradenitis suppurativa, Myositis, Multiple infected ulcers at distant sites, Infected burn wounds of a large area,
* Conditions requiring surgery that in and of itself would cure the infection or remove the infected site (eg, amputation)
* Conditions requiring emergent surgical intervention at the site of infection (eg, progressive necrotizing infections)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2008-09; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Atkin, Study Director — AstraZeneca; Zhang Yingyuan, Prof., Principal Investigator — Antibiotics Institute, Huashan Hospital Affilicated to Fudan University
Locations (13):
- China (13):
  - Research Site, Beijing, Beijing Municipality
  - Research Site, Guangzhou, Guangdong
  - Research Site, Wuhan, Hubei
  - Research Site, Changsha, Hunan
  - Research Site, Nanjing, Jiangsu
  - Research Site, Suzhou, Jiangsu
  - Research Site, Shenyang, Liaoning
  - Research Site, Shanghai, Shanghai Municipality
  - Research Site, Chengdu, Sichuan
  - Research Site, Chongqing
  - Research Site, Dalian
  - Research Site, Hangzhou
  - Research Site, Qingdao

REFERENCES:
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=300&filename=CSR-D1790C00003.pdf
- See also: CSR-D1790C00003.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=300&filename=CSR-D1790C00003.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 265 patients were randomised (daptomycin: 131 patients, comparator: 134 patients), with 264 patients receiving study treatment
Groups:
- Daptomycin: daptomycin 4mg/kg iv every 24hours
- Vancomycin, or Vancomycin Switch to Cloxacillin: vancomycin 1g per 12 hours, for 7-14 days; or switch to cloxacillin: 1 g every 6 hours or 2 g every 8 hours
Period: Overall Study
Arm/Group | Daptomycin | Vancomycin, or Vancomycin Switch to Cloxacillin
Started | 131 | 134
Completed | 111 | 110
Not Completed | 20 | 24
Not completed — Withdrawal by Subject | 9 | 5
Not completed — Physician Decision | 4 | 8
Not completed — Lost to Follow-up | 2 | 4
Not completed — incorrect enrolment | 3 | 4
Not completed — Protocol Violation | 0 | 1
Not completed — all others | 2 | 2

BASELINE CHARACTERISTICS:
Population: One patient was randomized but did not receive any study drug, so the patient was not included in FAS(full analysis set) population analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Daptomycin | Vancomycin, or Vancomycin Switch to Cloxacillin | Total
Number analyzed (Participants) | 130 | 134 | 264
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.2 (15.77) | 44.5 (16.02) | 44.3 (15.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 95 | 185
  Male | 40 | 39 | 79

OUTCOME MEASURES:

1. Primary Outcome: Change of Erythrocyte Volume Fraction(Percentage of Erythrocyte Volume in Total Volume of Blood)
Description: Erythrocyte volume fraction means under certain conditions, after centrifugation pressing, the percentage of erythrocyte volume in the total volume of blood
Time Frame: baseline to TOC(test of cure), for up to 4 weeks
Population: Only patients who had measurements in both baseline and TOC visit were included for the analysis. Change=TOC visit-baseline
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Daptomycin | Vancomycin, or Vancomycin Switch to Cloxacillin
Number analyzed (Participants) | 88 | 94
percentage | 0.00 (0.080) | 0.01 (0.033)

2. Primary Outcome: Change in Creatinine Clearance
Time Frame: baseline to TOC(test of cure), for up to 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ml/min
Arm/Group | Daptomycin | Vancomycin, or Vancomycin Switch to Cloxacillin
Number analyzed (Participants) | 80 | 79
ml/min | 9.91 (76.851) | 0.99 (21.232)

3. Primary Outcome: Change in Serum Total Creatine Phosphokinase (CPK)
Time Frame: baseline to TOC(test of cure), for up to 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Daptomycin | Vancomycin, or Vancomycin Switch to Cloxacillin
Number analyzed (Participants) | 77 | 83
IU/L | 0.60 (56.89) | -2.40 (46.05)

4. Primary Outcome: Change in Urine pH
Time Frame: baseline to TOC(test of cure), for up to 4 weeks
Population: Only patients who had measurements were included in the summary of a specific parameter at a specific time point. Change = TOC visit - baseline
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Daptomycin | Vancomycin, or Vancomycin Switch to Cloxacillin
Number analyzed (Participants) | 70 | 79
pH | -0.19 (0.960) | -0.30 (0.952)

5. Primary Outcome: Shift in ECG
Description: percentage of patients who were primarily tested as normal ECG at baseline and changed into abnormal ECG at TOC visit in all the patients with normal ECG at baseline
Time Frame: baseline to TOC(test of cure), for up to 4 weeks
Population: Only patients who had both measurements at baseline and TOC visit and those who got normal ECG resluts at baseline were included in the summary. Change=TOC visit-baseline
Measure: Number; unit: percentage of patients
Groups:
- Vancomycin, or Vancomycin Switch to Cloxacillin: vancomycin 1g per 12 hrs, for 7-14 days; or switch to cloxacillin: 1 g every 6 hours or 2 g every 8 hours
Arm/Group | Daptomycin | Vancomycin, or Vancomycin Switch to Cloxacillin
Number analyzed (Participants) | 56 | 51
percentage of patients | 5.4 | 7.8

6. Secondary Outcome: Blinded Investigator's Assessement of Clinical Response at TOC(Test of Cure)
Description: The percentage of patients who were cured or clinically improved in the clinical evaluable (CE) population of each arm at TOC visit was analyzed. CE population includes all the patients with no significant deviation from study protocol in full analysis set population, and meetting the following specific criteria: 1.receiving randomly dispensed study treatment at appropriate time(with a compliance of at least 80% or 4 days [3 days for patients evaluated as treatment failure]). 2.without the administration of potentially confounding non-investigational antibiotics (using one potentially effective non-investigational antibiotic for the treatment of primary infection due to other reasons than lack of efficacy from Day 1 to TOC [for systemicadministration of non-glycopeptides, >1 calendar day]). 3.meeting the study inclusion/exclusion criteria 4.necessary clinical evaluation performed (evaluation for effectiveness at TOC visit, except for the condition confirmed as clinically ineffective)
Time Frame: baseline and TOC, for up to 4 weeks
Population: There were 107 patients in daptomycin arm and 101 patients in comparator arm meeting the criteria of CE population and completed TOC visit.
Measure: Number; unit: percentage of patients
Arm/Group | Daptomycin | Vancomycin, or Vancomycin Switch to Cloxacillin
Number analyzed (Participants) | 107 | 101
percentage of patients | 93.5 | 90.1

7. Secondary Outcome: Blinded Investigator's Assessement of Clinical Response at EOT(End of Therapy)
Description: The percentage of patients who were cured or clinically improved in the clinical evaluable (CE) population at EOT visit was analyzed. CE population includes all the patients with no significant deviation from study protocol in full analysis set population, and meetting the following specific criteria: 1.receiving randomly dispensed study treatment at appropriate time(with a compliance of at least 80% or 4 days [3 days for patients evaluated as treatment failure]). 2.without the administration of potentially confounding non-investigational antibiotics (using one potentially effective non-investigational antibiotic for the treatment of primary infection due to other reasons than lack of efficacy from Day 1 to TOC [for systemicadministration of non-glycopeptides, >1 calendar day]). 3.meeting the study inclusion/exclusion criteria 4.necessary clinical evaluation performed (evaluation for effectiveness at TOC visit, except for the condition confirmed as clinically ineffective)
Time Frame: baseline and EOT(end of therapy), for up to 2 weeks
Population: There were 110 patients in daptomycin arm and 103 patients in comparator arm who both completed EOT visit and met the criteria of CE population
Measure: Number; unit: Percentage of patients
Arm/Group | Daptomycin | Vancomycin, or Vancomycin Switch to Cloxacillin
Number analyzed (Participants) | 110 | 103
Percentage of patients | 90.9 | 91.3

8. Secondary Outcome: Microbiological Response at TOC(Test of Cure)
Description: The microbiological response rate (removal or presumed removal) in ME(microbiological evaluable) population of daptomycin group and comparator group at TOC visit was analyzed. ME population includes all the patients with Gram-positive pathogenic bacteria isolated at baseline in CE population. Microbiological response rate means the percentage of strains which were removed or presumably removed at TOC visit in all the strains isolated from ME population at baseline.
Time Frame: baseline and TOC, for up to 4 weeks
Population: ME population includes all the patients with Gram-positive pathogenic bacteria isolated at baseline in CE population. There were 83 strains isolated from ME population of daptomycin arm(78 patients) and 86 strains from ME population in comparator arm(79 patients).
Measure: Number; unit: Percentage of strains
Units Other Than Participants: strains
Arm/Group | Daptomycin | Vancomycin, or Vancomycin Switch to Cloxacillin
Number analyzed (Participants) | 78 | 79
Number analyzed (strains) | 83 | 86
Percentage of strains | 94.0 | 90.7

9. Secondary Outcome: Microbiological Response at EOT(End of Therapy)
Description: The microbiological response rate (removal or presumed removal) in ME(microbiological evaluable) population of daptomycin group and comparator group at EOT visit was analyzed. ME population includes all the patients with Gram-positive pathogenic bacteria isolated at baseline in CE population. Microbiological response rate means the percentage of strains which were removed or presumably removed at EOT visit in all the strains isolated from ME population at baseline.
Time Frame: baseline and EOT, for up to 2 weeks
Population: ME population includes all the patients with Gram-positive pathogenic bacteria isolated at baseline in CE population. There were 86 strains isolated from 81 patients in daptomycin arm and 88 strains from 81 patients in comparator arm who met the criteria of ME population at EOT visit.
Measure: Number; unit: Percentage of strains
Units Other Than Participants: strains
Arm/Group | Daptomycin | Vancomycin, or Vancomycin Switch to Cloxacillin
Number analyzed (Participants) | 81 | 81
Number analyzed (strains) | 86 | 88
Percentage of strains | 89.5 | 87.5

10. Secondary Outcome: Per-pathogen(Methicillin Resistant Staphylococcus Aureus) Clinical Response at TOC(Test of Cure)
Description: This is the comparison of clinical efficacy by methicillin resistant staphylococcus aureus(MRSA) between the two groups. As the analysis was performed by specific pathogen in ME population and clinical efficacy was compared meanwhile, the clinical evaluation was based on the number of cases under the category of specific pathogen rather than the number of strains. Percentage of patients who were cured or improved at TOC visit in the patients who were identified with MRSA infection at baseline of both groups.
Time Frame: baseline and TOC, for up to 4 weeks
Population: There were 14 patients indentified MRSA infection in daptomycin group and 10 patients indentified with MRSA in comparator group.
Measure: Number; unit: Percentage of patients
Arm/Group | Daptomycin | Vancomycin, or Vancomycin Switch to Cloxacillin
Number analyzed (Participants) | 14 | 10
Percentage of patients | 100 | 90

11. Secondary Outcome: Per-pathogen(Methicillin Sensitive Staphylococcus Aureus) Clinical Response at TOC
Description: This is the comparison of clinical efficacy by methicillin sensitive staphylococcus aureus(MSSA) between the two groups. As the analysis was performed by specific pathogen in ME population and clinical efficacy was compared meanwhile, the clinical evaluation was based on the number of cases under the category of specific pathogen rather than the number of strains. Percentage of patients who were cured or improved at TOC visit in the patients who were identified with MSSA infection at baseline of both groups.
Time Frame: baseline and TOC(test of cure), for up to 4 weeks
Population: There were 33 patients indentified MSSA infection in daptomycin group and 37 patients indentified with MSSA in comparator group.
Measure: Number; unit: Percentage of patients
Arm/Group | Daptomycin | Vancomycin, or Vancomycin Switch to Cloxacillin
Number analyzed (Participants) | 33 | 37
Percentage of patients | 90.9 | 89.2

12. Secondary Outcome: Per-pathogen(Staphylococcus Aureus) Microbiological Response at TOC
Description: This is the comparison of clinical efficacy by staphylococcus aureus between the two groups. As the analysis was performed by specific pathogen in ME population and clinical efficacy was compared meanwhile, the clinical evaluation was based on the number of cases under the category of specific pathogen rather than the number of strains. Percentage of patients who were cured or improved at TOC visit in the patients who were identified with staphylococcus aureus infection at baseline of both groups.
Time Frame: baseline and TOC(test of cure), for up to 4 weeks
Population: There were 48 patients indentified staphylococcus aureus infection both in daptomycin group and in comparator group.
Measure: Number; unit: Percentage of patients
Arm/Group | Daptomycin | Vancomycin, or Vancomycin Switch to Cloxacillin
Number analyzed (Participants) | 48 | 48
Percentage of patients | 91.7 | 87.5

ADVERSE EVENTS:
Arm/Group | Daptomycin | Vancomycin, or Vancomycin Switch to Cloxacillin
Serious Adverse Events (participants affected / at risk) | 1 | 3
Other Adverse Events (participants affected / at risk) | 30 | 39
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Daptomycin | Vancomycin, or Vancomycin Switch to Cloxacillin
Pneumonia (Infections and infestations) | 1/131 (1) | 0/133 (0)
lung infection (Infections and infestations) | 0/131 (0) | 1/133 (1)
tuberculosis (Infections and infestations) | 0/131 (0) | 1/133 (1)
Hepatic Cirrhosis (Hepatobiliary disorders) | 0/131 (0) | 1/133 (1)
renal failure chronic (Renal and urinary disorders) | 0/131 (0) | 1/133 (1)
OTHER ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Daptomycin | Vancomycin, or Vancomycin Switch to Cloxacillin
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 7/131 (7) | 7/133 (7)
Aspartate Aminotransferase Increased (Investigations) | 6/131 (6) | 6/133 (6)
Blood Creatine Phosphokinase Increased (Investigations) | 4/131 (4) | 0/133 (0)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 1/131 (1) | 2/133 (2)
Blood Lactate Dehydrogenase Increased (Investigations) | 1/131 (1) | 1/133 (1)
RED BLOOD CELLS URINE POSITIVE (Investigations) | 1/131 (1) | 1/133 (1)
Blood Alkaline Phosphatase Increased (Investigations) | 0/131 (0) | 1/133 (1)
BLOOD CREATININE INCREASED (Investigations) | 0/131 (0) | 1/133 (1)
Blood Potassium Decreased (Investigations) | 0/131 (0) | 2/133 (2)
Blood Urine Present (Investigations) | 1/131 (1) | 0/133 (0)
ELECTROCARDIOGRAM QRS COMPLEX PROLONGE0D (Investigations) | 1/131 (1) | 0/133 (0)
Electrocardiogram T Wave Abnormal (Investigations) | 1/131 (1) | 0/133 (0)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0/131 (0) | 1/133 (1)
Monocyte Percentage Increased (Investigations) | 0/131 (0) | 1/133 (1)
Platelet Count Decreased (Investigations) | 0/131 (0) | 1/133 (1)
WHITE BLOOD CELLS URINE POSITIVE (Investigations) | 1/131 (1) | 0/133 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 0/131 (0) | 3/133 (5)
Rash (Skin and subcutaneous tissue disorders) | 1/131 (2) | 2/133 (7)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3/131 (3) | 2/133 (2)
Lung Infection (Infections and infestations) | 0/131 (0) | 1/133 (1)
PNEUMONIA (Infections and infestations) | 1/131 (1) | 0/133 (0)
Tuberculosis (Infections and infestations) | 0/131 (0) | 1/133 (1)
PYREXIA (General disorders) | 2/131 (2) | 1/133 (1)
CHEST DISCOMFORT (General disorders) | 1/131 (1) | 0/133 (0)
CHILLS (General disorders) | 0/131 (0) | 1/133 (1)
INJECTION SITE PAIN (General disorders) | 0/131 (0) | 1/133 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0/131 (0) | 2/133 (2)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1/131 (1) | 1/133 (1)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1/131 (1) | 0/133 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0/131 (0) | 1/133 (1)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 2/131 (2) | 0/133 (0)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 0/131 (0) | 1/133 (1)
ASCITES (Gastrointestinal disorders) | 0/131 (0) | 1/133 (1)
CONSTIPATION (Gastrointestinal disorders) | 1/131 (1) | 0/133 (0)
NAUSEA (Gastrointestinal disorders) | 0/131 (0) | 1/133 (1)
ANOREXIA (Metabolism and nutrition disorders) | 0/131 (0) | 1/133 (1)
AMNESIA (Nervous system disorders) | 0/131 (0) | 1/133 (1)
Dizziness (Nervous system disorders) | 0/131 (0) | 1/133 (1)
HEADACHE (Nervous system disorders) | 0/131 (0) | 1/133 (1)
MUSCLE CONTRACTIONS INVOLUNTARY (Nervous system disorders) | 1/131 (1) | 0/133 (0)
ANGINA PECTORIS (Cardiac disorders) | 1/131 (1) | 0/133 (0)
LEFT VENTRICULAR HYPERTROPHY (Cardiac disorders) | 0/131 (0) | 1/133 (1)
SUPRAVENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 0/131 (0) | 1/133 (1)
VENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 1/131 (1) | 0/133 (0)
DYSURIA (Renal and urinary disorders) | 1/131 (1) | 0/133 (0)
HAEMATURIA (Renal and urinary disorders) | 1/131 (1) | 0/133 (0)
RENAL FAILURE CHRONIC (Renal and urinary disorders) | 0/131 (0) | 1/133 (1)
Flushing (Vascular disorders) | 0/131 (0) | 2/133 (3)
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 0/131 (0) | 1/133 (1)
Insomnia (Psychiatric disorders) | 1/131 (1) | 0/133 (0)
PRURITUS GENITAL (Reproductive system and breast disorders) | 1/131 (1) | 0/133 (0)
BLOOD PHOSPHORUS INCREASED (Investigations) | 1/131 (1) | 0/133 (0) — BLOOD PHOSPHORUS INCREASED
BLOOD POTASSIUM INCREASED (Investigations) | 1/131 (1) | 0/133 (0)
BLOOD URIC ACID INCREASED (Investigations) | 1/131 (1) | 0/133 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other